CLINICAL TRIAL: NCT01465451
Title: A Prospective,Single-center,Randomized,Controlled Phase III Clinical Study Comparing Efficacy and Safety of Intraoperative Chemotherapy With 5-Fluorouracil Plus Curative Resection Versus Surgery Alone for Patients With Colorectal Cancer
Brief Title: Intra-operative Chemotherapy With 5-FU for Colorectal Cancer Patients Receiving Curative Resection: Efficacy and Safety
Acronym: IOCCRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHI-ZHONG PAN, Professor, Director, M.D., Ph.D, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSU 5010-2010016 IOCCRC
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; curative resection; intra-operative chemotherapy; 5-fluorouracil; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A- surgery alone (Active Comparator): all cases will receive standard surgical procedures of curative resection for colorectal cancer, without intra-operative chemotherapy.
  Interventions: Procedure: curative resection for colorectal cancer
- ARM B surgery plus chemotherapy (Experimental): all cases will receive standard surgical procedures described as arm A. In addition, all cases will receive 5-FU chemotherapy during operation.
  Interventions: Procedure: curative resection for colorectal cancer; Drug: intra-operative 5-FU chemotherapy

INTERVENTIONS:
Procedure: curative resection for colorectal cancer — right hemicolectomy for right colon cancer, transverse colectomy for transverse colon cancer, left hemicolectomy for left colon cancer, sigmoid colectomy for sigmoid colon cancer, and anterior resection or abdominal-perineal resection for rectal cancer.
  Other Names: curative resection for colorectal cancer.
Drug: intra-operative 5-FU chemotherapy — 5-FU, 1000 mg/m2, injection into bowel lumen at the beginning of resection 5-FU, 200 mg/m2, injection into portal vein via mesentery vein at the end of tumor removal and bowel reconstruction.
  5-FU, 300 mg/m2, left in abdominal cavity before incision closure. surgical procedures will be the same as described in ARM A.
  Other Names: intra-operative 5-FU chemotherapy for colorectal cancer
  Arms: ARM B surgery plus chemotherapy

SUMMARY:
The purpose of this study is to investigate efficacy and safety of intra-operative chemotherapy with 5-FU for colorectal cancer patients receiving curative resection. The hypothesis is intra-operative intervention might be the best timing for cancer cells killing by cytotoxic agents, when most of residual cancer cells may get a rapid growth after tumor debulking and may become more chemotherapy-sensitive. A three-step procedure is designed for intra-operative chemotherapy with 5-FU of 1500 mg/m2, including step 1 of intraluminal 5-FU injection with 1000 mg/m2 at beginning of resection, step 2 of 200mg/m2 5-FU injection into portal vein system via mesentery vein after tumor removal and finish of bowel reconstruction, and step 3 of 300mg/m2 5-FU left into the abdominal cavity before incision closure. The controlled arm receive curative resection only. All the other treatments will stick to the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed as adenocarcinoma of colon and rectum
* age 18-75 years
* eligible for curative surgical resection
* performance score: ECOG 0-1
* normal blood cells counts: WBC ≥ 4.0×10*9/L，PLT ≥ 100×10*9/L
* normal blood chemistry test: ALT/AST ≤ 2.5 ULN, TBil ≤ 1.5 ULN, BUN ≤ 1.5 ULN,Cr ≤ 1.5 ULN
* normal ECG
* no history of other malignant tumors
* no concomitant anti-cancer therapy

Exclusion Criteria:

* clinical bowel obstruction
* anticipated into another clinical trial within three months
* uncontrolled infection, serious internal medical diseases
* Pregnant or lactating women
* mentally abnormal patients
* patients known allergic to 5-FU

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2011-03; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 years
  3 years survival of recurrence-free, metastasisi-free, death-free after randomization.

SECONDARY OUTCOMES:
disease-free survival | 5 years
  5 years survival of recurrence-free, metastasis-free, and death-free survival after randomization.
safety profiles | 28 days after randomization
  complete blood cells counts, blood chemistry testing, all 28-day mortality after operation, all surgery-related complications

CONTACTS AND LOCATIONS:
Overall Officials: zhizhong pan, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Colorectal Surgery, 14Th Floor, Main Building, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang RX, Lin JZ, Lei J, Chen G, Li LR, Lu ZH, Ding PR, Huang JQ, Kong LH, Wang FL, Li C, Jiang W, Ke CF, Zhou WH, Fan WH, Liu Q, Wan DS, Wu XJ, Pan ZZ. Safety of intraoperative chemotherapy with 5-FU for colorectal cancer patients receiving curative resection: a randomized, multicenter, prospective, phase III IOCCRC trial (IOCCRC). J Cancer Res Clin Oncol. 2017 Dec;143(12):2581-2593. doi: 10.1007/s00432-017-2489-0. Epub 2017 Aug 28. PMID 28849265